CLINICAL TRIAL: NCT04054635
Title: A Randomized Clinical Trial of Silver Diamine Fluoride to Arrest Early Childhood Caries in Young Children
Brief Title: A Clinical Trial of Silver Diamine Fluoride to Arrest Early Childhood Caries in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Children's Hospital Research Institute of Manitoba (Other)
Responsible Party: Principal Investigator, Robert Schroth, DMD, MSc, PhD, Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019:068
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Early Childhood Caries
Keywords: silver diamine fluoride; randomized clinical trial; early childhood caries; severe early childhood caries; oral microbiome; treatment; arrest; application; frequency; regimen; cariogenic bacteria; early childhood oral health impact scale; oral health-related quality of of life; caries; oral bacteriome; oral mycobiome; cavitated lesions
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three application regimens of silver diamine fluoride (SDF) to cavitated caries lesions in primary teeth during the duration of the study. Regimen 1 will be two applications of SDF four months apart. Regimen 2 will be two applications of SDF six months apart. Regimen 3 will be two applications of SDF one month apart.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Regimen 1 (Experimental): Two applications of silver diamine fluoride (SDF) four months apart, which is the protocol frequency adopted by the Winnipeg Regional Health Authority's (WRHA) Clinical Guideline on SDF.
  Interventions: Device: Silver diamine fluoride
- Regimen 2 (Experimental): Two applications of silver diamine fluoride (SDF) six months apart, which is the American Dental Association's recommendation for SDF.
  Interventions: Device: Silver diamine fluoride
- Regimen 3 (Experimental): Two applications of silver diamine fluoride (SDF) one month apart, which is proposed in the American Academy of Pediatric Dentistry's clinical practice guidelines.
  Interventions: Device: Silver diamine fluoride

INTERVENTIONS:
Device: Silver diamine fluoride — Antibiotic liquid with anti-caries effects. A non-restorative option to manage cavitated caries lesions. Approved for clinical use in Canada in 2017.
  Other Names: Advantage Arrest Silver Diamine Fluoride 38%

SUMMARY:
Silver diamine fluoride (SDF) is an antibiotic liquid that has the potential to arrest Early Childhood Caries in young children and delay treatment until children can be seen in outpatient settings. While SDF received approval for clinical use in Canada in 2017 (i.e. Advantage Arrest TM/38% SDF), there has been little guidance on the frequency and duration of applications. This study evaluates the use of SDF at different frequencies to manage dental caries in young children. Potential oral microbiome changes in children receiving SDF treatments are also studied. The investigators hypothesize that two applications of SDF at different frequencies will yield similar arrest rates, and that SDF negatively influences the population of cariogenic bacteria in the oral microbiome. The investigators propose a randomized clinical trial to study the use of SDF to arrest cavitated lesions in primary teeth at different application regimens. Regimen 1 will be two applications of SDF four months apart. Regimen 2 will be two applications of SDF six months apart. Regimen 3 will be two applications of SDF one month apart. Arrest of caries lesions will be determined by assessing clinical hardness, colour change and size of lesions at baseline, at second visit, and at the final study visit. Children < 72 months of age with active caries will be recruited from community-based dental clinics or who are currently on a wait list for dental surgery under general anesthesia in Winnipeg, Manitoba. SDF will be applied on the day of recruitment to cavitated lesions involving dentin followed by 5%NaFV. Depending on which frequency regimen children are randomized to, participants will return for a second visit. At the second visit, caries lesions treated with SDF at baseline will be assessed to see if caries is arrested. A second application of SDF will be applied to these initially treated caries lesions followed by 5%NaFV. Participants will return for a third and final study visit according to the schedule of their randomized grouping. Caries lesions previously treated by SDF will be assessed once again. To investigate SDF's influence on the human oral microbiome, children from each regimen will have plaque samples collected. Samples will be obtained prior to SDF application at baseline, at the first follow-up visit, and at the final visit. Following nucleic acid isolation from plaque samples and amplicon sequencing, data analysis will be performed in lab using established methods.

DETAILED DESCRIPTION:
Good oral health during early childhood sets the foundation for a lifetime of optimal dental health. Unfortunately, many Canadian children develop Early Childhood Caries (ECC), defined as caries in the primary dentition in those < 72 months of age. ECC is a significant concern as not only can it increase the risk for caries throughout childhood and adolescence, but severe forms can impact health and well-being. Many with ECC suffer from an aggressive subtype, called severe ECC (S-ECC), which frequently requires rehabilitative dental surgery under general anesthesia (GA).

There is an urgent need to implement public health strategies to reduce the proportion of children developing ECC, especially S-ECC, and to manage effectively children who already have the disease. The challenge is that there are few effective interventions. Traditional primary prevention modalities have had little impact on reducing the incidence and severity of ECC in North America. Until recently there have been no effective non-surgical products for secondary prevention available. Though primary prevention is always preferred, secondary prevention can reduce the morbidity from caries and preserve the function of affected teeth until exfoliation.

Recent reports highlight the anti-caries effects of silver diamine fluoride (SDF). One systematic review and meta-analysis reported that 38% SDF is safe and effective in arresting dentin caries in primary teeth resulting in the arrest of 81% of active caries lesions. The recent American Dental Association (ADA) report on non-restorative management of caries prioritizes the use of SDF over other products to manage cavitated caries lesions. Despite this evidence, true consensus on the frequency of SDF applications in children with ECC is lacking. Further, the current American Academy of Pediatric Dentistry (AAPD) Clinical Practice Guidelines on SDF emphasize that research is needed on the use of SDF to arrest caries lesions in both primary and permanent teeth, specifically urging researchers to undertake randomized clinical trials (RCTs). SDF has the potential to arrest ECC in young children and delay treatment until children can be seen in outpatient settings, thereby reducing the need for rehabilitative dental surgery under GA.

While Advantage Arrest TM (38% SDF) received approval for clinical use in Canada in 2017, there has been little guidance on the frequency and duration of applications. Some proposed SDF protocols may not easily translate into dental public health clinical settings or work well in remote Indigenous communities, where access to care is often limited. Recommendations for frequent reapplication are not practical or realistic in these programs or remote regions where follow-up visits may be several months away and not within a matter of weeks. Since there was no clear protocol for dental professionals to follow for arresting caries in young children when SDF was approved for use in Canada in 2017, The investigators undertook a mixed-methods pilot feasibility study of SDF. Data from 40 children 40.2 ± 14.9 months of age are encouraging. Children with 239 active caries lesions in primary teeth underwent treatment with 38% SDF (followed by 5% sodium fluoride varnish/5%NaFV) at baseline and 4 months later. Treated lesions were assessed 4 and 8 months after baseline to determine arrest. The early childhood oral health impact scale (ECOHIS) questionnaire was completed at second and third visits to assess oral health related quality of life (OHRQoL). ECOHIS is a validated tool for use with parents/caregivers of children < 72 months of age. Arrest rates after one and two applications of SDF were 74.1% and 96.2%, respectively. OHRQoL was not found to be adversely affected by the success of SDF treatment. From these pilot data the investigators concluded that SDF is a promising agent to manage ECC, but at least two applications are recommended.

The purpose of this current study is to investigate the effectiveness of using SDF to arrest ECC in very young children randomized to different application frequency regimens. The investigators will also study potential oral microbiome changes in children receiving SDF treatment. The investigators hypothesize that two applications of SDF at different frequencies will yield similar arrest rates, and that SDF will negatively influence the population of cariogenic bacteria in the oral microbiome.

The investigators propose a RCT to study the use of SDF to arrest cavitated caries lesions in primary teeth at different application regimens. This study is novel, as this would be the first RCT of SDF conducted in Canada. Regimen 1 will be two applications of SDF four months apart, which is the protocol frequency adopted by the Winnipeg Regional Health Authority's (WRHA) Clinical Guideline on SDF. Regimen 2 will be two applications of SDF six months apart (ADA recommendation). Regimen 3 will be two applications of SDF one month apart, which is proposed in the AAPD's clinical practice guideline. The ADA recently indicated that SDF should be prioritized over 5%NaFV for non-restorative management of cavitated lesions. Thus, a control group receiving solely fluoride varnish will not be included as this would now be considered unethical and substandard care. However, the investigators will attempt to follow as a comparison group those children whose parents/caregivers do not consent to SDF to manage their child's caries and only choose 5%NaFV.

Arrest of caries lesions will be determined by assessing clinical hardness, colour change, and size of lesions at baseline, at second visit, and at the final study visit. Children will be recruited over eight months. The investigators will perform block randomization by site in order to achieve equal proportions in each regimen by clinic site of recruitment. Following informed consent the child's parent/caregiver will complete a short questionnaire (via interview) on general and dental health, oral hygiene, dietary intake of sugars, and family demographics along with the ECOHIS to assess OHRQL. SDF will be applied on the day of recruitment to cavitated lesions involving dentin followed by 5%NaFV. Depending on which frequency regimen children are randomized to, participants will return for a second visit. During this second visit, caries lesions treated with SDF at baseline will be assessed to see if caries is arrested as determined through measures of hardness, colour change, and size. At this same visit a second application of SDF will be applied to these initially treated caries lesions followed by 5%NaFV. Children and parents will return for the third and final study visit according to the schedule of their randomized grouping. Parents/caregivers will complete a follow-up questionnaire similar to the baseline tool. Caries lesions previously treated by SDF will be assessed for clinical hardness, colour change and size to determine if they have arrested.

As ECC is age specific, participants will be < 72 months of age with active caries and their parents/caregivers. The majority will be recruited from community-based dental clinics in Winnipeg or who are currently on a wait list for dental surgery under GA in Winnipeg. The investigators found that these were ideal sites for the recently completed feasibility trial of SDF. Participation will be restricted to children living in the Winnipeg region or within a one hour drive of Winnipeg to minimize the risk of loss-to-follow-up. Eligibility criteria are designed to select young children who have active caries, and thus are at an increased risk of morbidity from existing caries and onset of new caries.

Sample size for this pilot study has been determined in discussion with a collaborator. The intent of the study is not to compare arrest rates between groups to see which yields higher and more significant arrest rates. Rather, the investigators are interested in determining whether the three different regimens will yield arrest rates within a range of what is determined to be clinically acceptable. Based on the recent pilot feasibility study of SDF with 40 children (with 239 lesions), the investigators reported an arrest rate of approximately 96% following two applications of SDF. Results from a recent systematic review state that 80% of lesions can arrest because of SDF. The investigators believe that a range of arrest rates from 80% to 96% yield similar beneficial outcomes in the clinical setting. Based on the pilot study, 40 children had 239 lesions (average 6 lesions/child). With the pilot sample of 239 lesions, it is possible to estimate an arrest rate with a 95% confidence interval to be accurate within ± 6.5%. With 400 lesions anticipated in the proposed recruitment sample, the 95% confidence interval for the arrest rate would be ± 5.0%. The investigators propose three SDF regimen groups and anticipate that each group will have 22 children anticipating an average of six lesions. This would mean 396 lesions would be followed in this study. The investigators anticipate that with 400 lesions the percent of arrest will be within ± 5% if 22 children are in each group. To deal with potential drop-outs and loss-to-follow-up of up to 20% the investigators will over recruit by 22.7% into each group and recruit 27 per group. The investigators anticipate the successful recruitment of 10 children each month.

Clinical outcomes assessed will include the proportion of lesions arrested (i.e., "arrest rate" = total number lesions arrested / total number of lesions treated), the number of children with arrested caries, and the number of children requiring dental surgery under GA. The investigators will also record dmft and dmfs scores for each child at baseline and at subsequent study visits. The dmft and dmfs scores are cumulative counts of the total number of primary teeth or surfaces decayed, missing due to, or filled because of caries.

Caries activity will be determined according to hardness and colour of the caries lesion. Hardness is the best indicator of dentinal tissue caries activity. The hardness of caries lesions will be assessed by applying light force to the lesion with a ball ended probe and by classifying the lesion into one of three hardness categories: 1) very soft; 2) medium; or 3) very hard. The investigators will record these ratings of hardness of lesions on the Clinical Record Forms at the baseline visit, second visit, and third (final) clinical visit. The Clinical Record Forms will be those used in the pilot feasibility study of SDF. The colour of caries lesions will also be assessed. Dentin colour of each caries lesion will be classified as: 1) yellow; 2) brown; or 3) black. The colour black is associated with arrested caries. The size of caries lesions will also be measured (in mm) at the baseline, second, and third clinical visits.

To investigate SDF's influence on the human oral microbiome, ten children from each regimen will have plaque samples collected. Samples will be obtained prior to SDF application at baseline, at the first follow-up visit, and at the final visit. Following nucleic acid isolation from plaque samples and amplicon sequencing, data analysis will be performed in lab using established methods.

Problems and adverse events will be recorded and reported to the University of Manitoba's ethics office.

ELIGIBILITY:
Inclusion Criteria:

1. Child is < 72 months of age with early childhood caries (ECC) with active lesions (International Caries Detection and Assessment System codes 5 or 6).
2. Child has ≥ 1 primary tooth with caries that is eligible to receive SDF. Eligible primary teeth must: a) have soft cavitated caries lesions extending into dentin; b) the cavitated lesions must allow for direct application of silver diamine fluoride (SDF). Teeth that meet any of the PUFA (pulpal involvement, ulceration, fistula, and abscess) index criteria (i.e. spontaneous pain due to caries, pulp exposure, mobility, signs of pulpal infection such as abscess, fistula, or swelling) will be excluded. However, a child would still be eligible even if they have at least one tooth that meets PUFA criteria, but other eligible teeth with caries do not.

Exclusion Criteria:

1. Child is allergic or has a sensitivity to silver or other heavy metal ions.
2. Child has hereditary generalized developmental defects of enamel (e.g. Amelogenesis Imperfecta, Dentinogenesis Imperfecta)
3. Child has severe medical problems that limit participation.
4. Child requires immediate rehabilitation under general anesthesia (GA) because of severe infection or pain.
5. Antibiotic use within the last 2 weeks.

Max Age: 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Schroth, Principal Investigator — University of Manitoba
Locations (1):
- Children's Hospital Research Institute of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Policy on Early Childhood Caries (ECC): Classifications, Consequences, and Preventive Strategies. Pediatr Dent. 2017 Sep 15;39(6):59-61. No abstract available. PMID 29179321
- [Background] Schroth RJ, Levi JA, Sellers EA, Friel J, Kliewer E, Moffatt ME. Vitamin D status of children with severe early childhood caries: a case-control study. BMC Pediatr. 2013 Oct 25;13:174. doi: 10.1186/1471-2431-13-174. PMID 24160554
- [Background] Schroth RJ, Harrison RL, Moffatt ME. Oral health of indigenous children and the influence of early childhood caries on childhood health and well-being. Pediatr Clin North Am. 2009 Dec;56(6):1481-99. doi: 10.1016/j.pcl.2009.09.010. PMID 19962032
- [Background] Schroth RJ, Levi J, Kliewer E, Friel J, Moffatt ME. Association between iron status, iron deficiency anaemia, and severe early childhood caries: a case-control study. BMC Pediatr. 2013 Feb 7;13:22. doi: 10.1186/1471-2431-13-22. PMID 23388209
- [Background] Schroth RJ, Quinonez C, Shwart L, Wagar B. TREATING EARLY CHILDHOOD CARIES UNDER GENERAL ANESTHESIA: A NATIONAL REVIEW OF CANADIAN DATA. J Can Dent Assoc. 2016 Jul;82:g20. PMID 27548666
- [Background] Schroth RJ, Smith WF. A review of repeat general anesthesia for pediatric dental surgery in Alberta, Canada. Pediatr Dent. 2007 Nov-Dec;29(6):480-7. PMID 18254418
- [Background] Fisher-Owens SA, Gansky SA, Platt LJ, Weintraub JA, Soobader MJ, Bramlett MD, Newacheck PW. Influences on children's oral health: a conceptual model. Pediatrics. 2007 Sep;120(3):e510-20. doi: 10.1542/peds.2006-3084. PMID 17766495
- [Background] Selwitz RH, Ismail AI, Pitts NB. Dental caries. Lancet. 2007 Jan 6;369(9555):51-9. doi: 10.1016/S0140-6736(07)60031-2. PMID 17208642
- [Background] Peng JJ, Botelho MG, Matinlinna JP. Silver compounds used in dentistry for caries management: a review. J Dent. 2012 Jul;40(7):531-41. doi: 10.1016/j.jdent.2012.03.009. Epub 2012 Apr 3. PMID 22484380
- [Background] Chu CH, Lo EC, Lin HC. Effectiveness of silver diamine fluoride and sodium fluoride varnish in arresting dentin caries in Chinese pre-school children. J Dent Res. 2002 Nov;81(11):767-70. doi: 10.1177/0810767. PMID 12407092
- [Background] Rosenblatt A, Stamford TC, Niederman R. Silver diamine fluoride: a caries "silver-fluoride bullet". J Dent Res. 2009 Feb;88(2):116-25. doi: 10.1177/0022034508329406. PMID 19278981
- [Background] Horst JA, Ellenikiotis H, Milgrom PL. UCSF Protocol for Caries Arrest Using Silver Diamine Fluoride: Rationale, Indications and Consent. J Calif Dent Assoc. 2016 Jan;44(1):16-28. PMID 26897901
- [Background] Milgrom P, Horst JA, Ludwig S, Rothen M, Chaffee BW, Lyalina S, Pollard KS, DeRisi JL, Mancl L. Topical silver diamine fluoride for dental caries arrest in preschool children: A randomized controlled trial and microbiological analysis of caries associated microbes and resistance gene expression. J Dent. 2018 Jan;68:72-78. doi: 10.1016/j.jdent.2017.08.015. Epub 2017 Sep 1. PMID 28866468
- [Background] Gao SS, Zhao IS, Hiraishi N, Duangthip D, Mei ML, Lo ECM, Chu CH. Clinical Trials of Silver Diamine Fluoride in Arresting Caries among Children: A Systematic Review. JDR Clin Trans Res. 2016 Oct;1(3):201-210. doi: 10.1177/2380084416661474. Epub 2016 Aug 20. PMID 30931743
- [Background] Slayton RL, Urquhart O, Araujo MWB, Fontana M, Guzman-Armstrong S, Nascimento MM, Novy BB, Tinanoff N, Weyant RJ, Wolff MS, Young DA, Zero DT, Tampi MP, Pilcher L, Banfield L, Carrasco-Labra A. Evidence-based clinical practice guideline on nonrestorative treatments for carious lesions: A report from the American Dental Association. J Am Dent Assoc. 2018 Oct;149(10):837-849.e19. doi: 10.1016/j.adaj.2018.07.002. PMID 30261951
- [Background] Use of Silver Diamine Fluoride for Dental Caries Management in Children and Adolescents, Including Those with Special Health Care Needs. Pediatr Dent. 2017 Sep 15;39(6):146-155. PMID 29179353
- [Background] Horst JA. Silver Fluoride as a Treatment for Dental Caries. Adv Dent Res. 2018 Feb;29(1):135-140. doi: 10.1177/0022034517743750. PMID 29355428
- [Background] Pahel BT, Rozier RG, Slade GD. Parental perceptions of children's oral health: the Early Childhood Oral Health Impact Scale (ECOHIS). Health Qual Life Outcomes. 2007 Jan 30;5:6. doi: 10.1186/1477-7525-5-6. PMID 17263880
- [Background] Jankauskiene B, Virtanen JI, Kubilius R, Narbutaite J. Oral health-related quality of life after dental general anaesthesia treatment among children: a follow-up study. BMC Oral Health. 2014 Jul 1;14:81. doi: 10.1186/1472-6831-14-81. PMID 24984901
- [Background] Ward TL, Dominguez-Bello MG, Heisel T, Al-Ghalith G, Knights D, Gale CA. Development of the Human Mycobiome over the First Month of Life and across Body Sites. mSystems. 2018 Mar 6;3(3):e00140-17. doi: 10.1128/mSystems.00140-17. eCollection 2018 May-Jun. PMID 29546248
- [Background] Walters W, Hyde ER, Berg-Lyons D, Ackermann G, Humphrey G, Parada A, Gilbert JA, Jansson JK, Caporaso JG, Fuhrman JA, Apprill A, Knight R. Improved Bacterial 16S rRNA Gene (V4 and V4-5) and Fungal Internal Transcribed Spacer Marker Gene Primers for Microbial Community Surveys. mSystems. 2015 Dec 22;1(1):e00009-15. doi: 10.1128/mSystems.00009-15. eCollection 2016 Jan-Feb. PMID 27822518
- [Background] Usyk M, Zolnik CP, Patel H, Levi MH, Burk RD. Novel ITS1 Fungal Primers for Characterization of the Mycobiome. mSphere. 2017 Dec 13;2(6):e00488-17. doi: 10.1128/mSphere.00488-17. eCollection 2017 Nov-Dec. PMID 29242834
- [Background] Agnello M, Marques J, Cen L, Mittermuller B, Huang A, Chaichanasakul Tran N, Shi W, He X, Schroth RJ. Microbiome Associated with Severe Caries in Canadian First Nations Children. J Dent Res. 2017 Nov;96(12):1378-1385. doi: 10.1177/0022034517718819. Epub 2017 Jul 14. PMID 28709393
- [Background] Peters BA, Wu J, Hayes RB, Ahn J. The oral fungal mycobiome: characteristics and relation to periodontitis in a pilot study. BMC Microbiol. 2017 Jul 12;17(1):157. doi: 10.1186/s12866-017-1064-9. PMID 28701186
- [Background] Schroth RJ, Jeal NS, Kliewer E, Sellers EA. The relationship between vitamin D and severe early childhood caries: a pilot study. Int J Vitam Nutr Res. 2012 Feb;82(1):53-62. doi: 10.1024/0300-9831/a000094. PMID 22811377
- [Background] Davidson K, Schroth RJ, Levi JA, Yaffe AB, Mittermuller BA, Sellers EAC. Higher body mass index associated with severe early childhood caries. BMC Pediatr. 2016 Aug 20;16:137. doi: 10.1186/s12887-016-0679-6. PMID 27543009
- [Background] Prowse S, Schroth RJ, Wilson A, Edwards JM, Sarson J, Levi JA, Moffatt ME. Diversity considerations for promoting early childhood oral health: a pilot study. Int J Dent. 2014;2014:175084. doi: 10.1155/2014/175084. Epub 2014 Jan 30. PMID 24624141
- [Background] Schroth RJ, Edwards JM, Brothwell DJ, Yakiwchuk CA, Bertone MF, Mellon B, Ward J, Ellis M, Hai-Santiago K, Lawrence HP, Moffatt ME. Evaluating the impact of a community developed collaborative project for the prevention of early childhood caries: the Healthy Smile Happy Child project. Rural Remote Health. 2015 Oct-Dec;15(4):3566. Epub 2015 Nov 4. PMID 26530126
- [Background] Macintosh AC, Schroth RJ, Edwards J, Harms L, Mellon B, Moffatt M. The impact of community workshops on improving early childhood oral health knowledge. Pediatr Dent. 2010 Mar-Apr;32(2):110-7. PMID 20483013
- [Background] Schroth RJ, Moore P, Brothwell DJ. Prevalence of early childhood caries in 4 Manitoba communities. J Can Dent Assoc. 2005 Sep;71(8):567. PMID 16202195
- [Background] Schroth RJ, Wilson A, Prowse S, et al. Looking back to move forward: understanding service provider, parent, and caregiver views on early childhood oral health promotion in Manitoba, Canada. Can J Dent Hyg. 2014 Jan;48(3):99-108.
- [Background] Canadian Institute for Health Information. Treatment of Preventable Dental Cavities in Preschoolers: A Focus on Day Surgery Under General Anesthesia. Ottawa, ON: CIHI; 2013. p. 1-34.
- [Background] Sihra R, Schroth RJ, Bertone M, Martin H, Patterson B, Mittermuller BA, Lee V, Patterson B, Moffatt ME, Klus B, Fontana M, Robertson L. The Effectiveness of Silver Diamine Fluoride and Fluoride Varnish in Arresting Caries in Young Children and Associated Oral Health-Related Quality of Life. J Can Dent Assoc. 2020 Jun;86:k9. PMID 32543369
- [Background] Grant CG, Daymont C, Rodd C, Mittermuller BA, Pierce A, Kennedy T, Singh S, Moffatt MEK, Schroth RJ. Oral Health-Related Quality of Life of Canadian Preschoolers with Severe Caries After Dental Rehabilitation Under General Anesthesia. Pediatr Dent. 2019 May 15;41(3):221-228. PMID 31171075
- [Derived] Manerkar M, de Jesus VC, Mittermuller BA, Lee VHK, Singh S, Bertone M, Chelikani P, Schroth RJ. Effects of silver diamine fluoride on oral bacteriome and mycobiome: a randomized clinical trial. BMC Oral Health. 2025 Oct 21;25(1):1643. doi: 10.1186/s12903-025-06986-0. PMID 41120980
- [Derived] Schroth RJ, Bajwa S, Lee VHK, Mittermuller BA, Singh S, Cruz de Jesus V, Bertone M, Chelikani P. An open-label, parallel-group, randomized clinical trial of different silver diamine fluoride application intervals to arrest dental caries. BMC Oral Health. 2024 Sep 4;24(1):1036. doi: 10.1186/s12903-024-04791-9. PMID 39227897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants under 72 months of age with early childhood caries were recruited between October 2019 and June 2021 from community dental clinics in Winnipeg, Manitoba, Canada (Access Downtown, Mount Carmel Clinic, and SMILE Plus Children's Dental Clinic). Study visits took place at these clinics or at the Children's Hospital Research Institute of Manitoba.
Pre-assignment Details: Children were not approached if: caries were not ICDAS (international caries detection and assessment system) codes 5/6; affected teeth met PUFA (pulpal involvement, ulceration, fistula, and abscess) index criteria; children had allergy/sensitivity to silver/heavy metal ions, developmental defects of enamel, severe medical issues, used antibiotics within two weeks of recruitment, or required immediate rehabilitation under general anesthesia. Participants were randomized using sealed envelopes.
Period: First Visit (Baseline)
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Started | 28 | 28 | 28
Completed | 28 | 28 | 28
Not Completed | 0 | 0 | 0
Period: Second Visit (First Follow-up)
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Started | 28 | 28 | 28
Completed | 28 | 27 (Participants lost to follow-up were still in the study as a part of intention-to-treat analysis, where those lost to follow-up were still included (i.e., still 28 participants in regimen 2), and we acted as though there were no changes to the lesions of these participants at subsequent (missed) visits. This approach was chosen since it preserves randomization and was the best neutral response for the unknown status of lesions.) | 28
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Period: Third Visit (Second Follow-up)
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Started | 28 | 27 | 28
Completed | 27 (Participants lost to follow-up were still in the study as a part of intention-to-treat analysis, where those lost to follow-up were still included (i.e., still 28 participants in regimen 1), and we acted as though there were no changes to the lesions of these participants at subsequent (missed) visits. This approach was chosen since it preserves randomization and was the best neutral response for the unknown status of lesions.) | 27 | 28
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 | Total
Number analyzed (Participants) | 28 | 28 | 28 | 84
Age, Continuous [Mean (Standard Deviation); unit: months] | 40.5 (12.6) | 48.9 (14.2) | 43.9 (15.0) | 44.4 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 9 | 35
  Male | 13 | 17 | 19 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Background: African | 11 | 6 | 15 | 32
  Background: Asian | 7 | 12 | 5 | 24
  Background: European | 2 | 3 | 3 | 8
  Background: Indigenous | 8 | 7 | 5 | 20
Newcomer to Canada [Count of Participants; unit: Participants] | 4 | 5 | 5 | 14
Frequency of tooth brushing [Count of Participants; unit: Participants]
  Twice daily | 17 | 17 | 18 | 52
  Once daily | 8 | 10 | 6 | 24
  Less than once a day | 3 | 1 | 4 | 8
Use of fluoridated toothpaste [Count of Participants; unit: Participants]
  Yes | 24 | 22 | 23 | 69
  No | 1 | 2 | 3 | 6
  Do not know | 3 | 4 | 2 | 9
Has dental insurance [Count of Participants; unit: Participants] | 20 | 19 | 19 | 58
Has tooth pain [Count of Participants; unit: Participants] | 1 | 2 | 2 | 5
Total number of teeth treated [Number; unit: teeth] | 121 | 110 | 143 | 374
Total number of lesions treated [Number; unit: lesions] | 166 | 143 | 196 | 505
Mean number of teeth treated [Mean (Standard Deviation); unit: teeth] | 4.3 (3.1) | 7.6 (19.9) | 5.1 (2.7) | 4.6 (2.8)
Mean number of lesions treated [Mean (Standard Deviation); unit: lesions] | 5.9 (5.2) | 5.1 (4.1) | 7.0 (4.8) | 6.0 (4.7)
Mean dmft [Mean (Standard Deviation); unit: dmft index] — The dmft index represents the number of decayed, missing due to caries, and filled primary teeth. The total number of primary human teeth is 20; thus, the maximum dmft index is 20, and the minimum value is 0 (higher scores indicate poorer oral health and a greater number of decayed, missing due to caries, and filled primary teeth).
  dmft index | 6.2 (4.7) | 7.3 (4.1) | 7.0 (4.7) | 6.8 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Overall Arrest Rates
Description: Total number of lesions arrested/total number of lesions treated
Time Frame: 8 months, 12 months, and 2 months
Measure: Number; unit: percentage of lesions arrested
Units Other Than Participants: lesions
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Number analyzed (Participants) | 28 | 28 | 28
Number analyzed (lesions) | 166 | 143 | 196
percentage of lesions arrested
  Second visit (first follow-up) | 81.3 | 61.5 | 78.1
  Third visit (second follow-up) | 95.8 | 72.0 | 98.0

2. Primary Outcome: Anterior Teeth Arrest Rates
Description: Total number of anterior lesions arrested/total number of anterior lesions treated.
Time Frame: 8 months, 12 months, and 2 months
Measure: Number; unit: percentage of lesions arrested
Units Other Than Participants: lesions
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Number analyzed (Participants) | 28 | 28 | 28
Number analyzed (lesions) | 94 | 73 | 133
percentage of lesions arrested
  Second visit (first follow-up) | 83.0 | 75.3 | 85.0
  Third visit (second follow-up) | 97.9 | 74.0 | 99.2

3. Primary Outcome: Posterior Arrest Rates
Description: Total number of posterior lesions arrested/total number of posterior lesions treated.
Time Frame: 8 months, 12 months, and 2 months
Measure: Number; unit: percentage of lesions arrested
Units Other Than Participants: lesions
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Number analyzed (Participants) | 28 | 28 | 28
Number analyzed (lesions) | 72 | 70 | 63
percentage of lesions arrested
  Second visit (first follow-up) | 79.2 | 48.6 | 63.5
  Third visit (second follow-up) | 93.1 | 70.0 | 95.2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 21 months from October 2019 to June 2021. Depending on the participant's group, adverse events were monitored/assessed over three months, eight months, or 12 months (i.e., from recruitment/baseline to study completion).
Description: Because of the nature of early childhood caries in this study, there is no risk of death for participants; thus, all-cause mortality was not monitored/assessed. The inclusion criteria for the study and the treatment involved prevents any serious hospitalization of participants or any serious health risks.
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28

LIMITATIONS AND CAVEATS:
A limitation of this study is the significant difference in the number of teeth and lesions treated between the three groups. The six-month interval group (regimen 2) had a lower number of lesions treated than the one-month (regimen 3) or four-month (regimen 1) interval groups. Since arrest rates were analyzed using a pooled sample, the six-month interval group may have been disadvantaged from a lack of additional lesions to be examined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT04054635/Prot_SAP_000.pdf